CLINICAL TRIAL: NCT01500109
Title: Analgesic Efficacy of Oral Versus Intravenous Acetaminophen for Primary Pediatric Cleft Palate Repair; a Randomized, Double, Blinded, Placebo Controlled Study
Brief Title: Efficacy of Oral Versus Intravenous Acetaminophen for Primary Pediatric Cleft Palate Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5110257
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Cleft Palate
Keywords: cleft palate surgery; post-operative pain management; Acetaminophen
MeSH Terms: conditions — Cleft Palate | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ofirmev® (Experimental): Oral inert cherry syrup will be administered preoperatively as placebo for oral acetaminophen. Ofirmev® will be administered in the operating room once intravenous access is established. Patients will receive standardized dose of local anesthetic (Lidocaine 0.5% with Epinephrine) infiltration by the surgeon before surgical incision as well as at the completion of surgery with Bupivacaine 0.25% with Epinephrine. Postoperatively patients will receive Ofirmev® every 6 hours as well as placebo oral cherry elixir every 6 hours and morphine as needed for 24 hours.
  Interventions: Drug: Ofirmev®
- Oral acetaminophen (Active Comparator): Patients will receive oral acetaminophen cherry elixir preoperatively. After intravenous access is obtained intraoperatively patients will receive placebo for Ofirmev® (saline). Patients will receive standardized dose of local anesthetic (Lidocaine 0.5% with Epinephrine) infiltration by the surgeon prior to surgical incision as wel as at the completion of surgery with Bupivacaine 0.25% with Epinephrine. Postoperatively patient will receive oral acetaminophen every six hours and intravenous placebo (normal saline) for intravenous acetaminophen. Intravenous morphine will be administered as needed for 24 hours.
  Interventions: Drug: Oral acetaminophen
- Opioid only (Placebo Comparator): This group will receive placebo oral cherry elixir prior to going to the operating room and placebo Ofirmev® after securing intravenous access in the operating room with redosing every six hours. They will receive local anesthetic (Lidocaine 0.5% with Epinephrine) infiltration by the surgeon prior to incision as well as at the completion of surgery with Bupivicaine 0.25% with Epinephrine. Postoperatively they will receive only Morphine prn for pain control.
  Interventions: Drug: Opioid only

INTERVENTIONS:
Drug: Oral acetaminophen — Oral acetaminophen administered as a cherry flavored elixir will be dosed preoperatively 15 mg/kg and redosed every 6 hours for 24 hours. Placebo oral acetaminophen will be administered to the other two arms of the study according to the same timetable. Intraoperative opioids (Fentanyl or Morphine) will be administered as deemed necessary by anesthesia care team. in the PACU, fentanyl 0.5-1 mcg/kg will be administered for moderate-severe pain. Once discharged from PACU, morphine 0.05 mg/kg will be given every 3 hours as needed.
  Arms: Oral acetaminophen
Drug: Ofirmev® — Intravenous acetaminophen is initiated after intravenous access is obtained intraoperatively and before surgical incision. Dosing is age based as follows: 5 months-2 years 12.5 mg/kg, 2-5 years 15 mg/kg. Redosing will be every 6 hours for 24 hours. The two other arms will receive a placebo in the form of normal saline given intravenously. Intraoperative opioids will be administered as deemed necessary by anesthesia care team. in the PACU, fentanyl 0.5-1 mcg/kg will be administered for moderate-severe pain. Once discharged from PACU, morphine 0.05 mg/kg will be given every 3 hours as needed.
  Arms: Ofirmev®
Drug: Opioid only — Intraoperative opioids (Fentanyl or Morphine) will be administered as deemed necessary by anesthesia care team. in the PACU, fentanyl 0.5-1 mcg/kg will be administered for moderate-severe pain. Once discharged from PACU, morphine 0.05 mg/kg will be given every 3 hours as needed.
  Arms: Opioid only

SUMMARY:
The purpose of this investigator-initiated study is to determine whether acetaminophen is an effective pain reliever for primary cleft palate repair in children and possesses opioid sparing effects. Additionally, the investigators will determine if patients who receive acetaminophen have less opioid related side-effects. The study will have three study groups based on whether the patient receives Ofirmev® and opioids (Fentanyl and Morphine), oral acetaminophen elixir and opioids (Fentanyl and Morphine), or opioids (Fentanyl and Morphine) alone. Total opioid (Fentanyl and Morphine) consumption will be tracked for the intraoperative period and 24 hours after surgery for all patients within the study and converted to morphine equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Children 5 months to five years of age
* ASA physical status I or II
* primary cleft palate repair alone or in some combination with bilateral myringotomy with tympanostomy (BMT), alveoplasty, vomer flap, rhinoplasty, and or cleft lip repair.?

Exclusion Criteria:

* Repeat/revision cleft palate repair
* Contraindications to acetaminophen administration (liver or renal dysfunction, allergy)
* Chronic pain medications
* Diagnosis of chronic pain syndrome
* Contraindications to morphine (renal impairment, allergy)
* Seizure disorders and/or taking anti-seizure medications
* Contraindications to oral midazolam (liver dysfunction, allergy)
* Allergy to local anesthetics

Ages: 5 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelan Nour, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofirmev®: Oral inert cherry syrup will be administered preoperatively as placebo for oral acetaminophen. Ofirmev will be administered in the operating room once intravenous access is established. Patients will receive standardized dose of local anesthetic (Lidocaine 0.5% with Epinephrine) infiltration by the surgeon before surgical incision as well as at the completion of surgery with Bupivacaine 0.25% with Epinephrine. Postoperatively patients will receive Ofirmev® every 6 hours as well as placebo oral cherry elixir every 6 hours and morphine as needed for 24 hours.
  Ofirmev®: Intravenous acetaminophen is initiated after intravenous access is obtained intraoperatively and before surgical incision. Dosing is age based as follows: 5 months-2 years 12.5 mg/kg, 2-5 years 15 mg/kg. Redosing will be every 6 hours for 24 hours. The two other arms will receive a placebo in the form of normal saline given intravenously. Intraoperative opioids will be administered as deemed necessary by anesthesia c
- Oral Acetaminophen: Patients will receive oral acetaminophen cherry elixir preoperatively. After intravenous access is obtained intraoperatively patients will receive placebo for Ofirmev (saline). Patients will receive standardized dose of local anesthetic (Lidocaine 0.5% with Epinephrine) infiltration by the surgeon prior to surgical incision as wel as at the completion of surgery with Bupivacaine 0.25% with Epinephrine. Postoperatively patient will receive oral acetaminophen every six hours and intravenous placebo (normal saline) for intravenous acetaminophen. Intravenous morphine will be administered as needed for 24 hours.
  Oral acetaminophen: Oral acetaminophen administered as a cherry flavored elixir will be dosed preoperatively 15 mg/kg and redosed every 6 hours for 24 hours. Placebo oral acetaminophen will be administered to the other two arms of the study according to the same timetable. Intraoperative opioids (Fentanyl or Morphine) will be administered as deemed necessary by anesthesia care t
Period: Overall Study
Arm/Group | Ofirmev® | Oral Acetaminophen | Opioid Only
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI left institution without completing results. All efforts to contact PI for data have been unsuccessful. No data available to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofirmev® | Oral Acetaminophen | Opioid Only | Total
Number analyzed (Participants) | 15 | 14 | 16 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 14 | 16 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Months] | 7.7 [6.6 to 10.4] | 8.7 [7.0 to 11.7] | 8.2 [7.2 to 10.1] | 8.2 [6.6 to 11.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 10 | 23
  Male | 10 | 6 | 6 | 22
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Opioid (Fentanyl and Morphine) Consumption
Description: The primary outcome measure of the study will be to measure opioid (Fentanyl and Morphine) consumption during the intraoperative period first postoperative 24 hours (measured in morphine equivalents).
Time Frame: intraoperative period and first postoperative 24 hours
Population: as for baseline characteristics
Arm/Group | Ofirmev® | Oral Acetaminophen | Opioid Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: PI left institution without completing results. All efforts to contact PI for data have been unsuccessful. No data available to report.
Arm/Group | Ofirmev® | Oral Acetaminophen | Opioid Only
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes